CLINICAL TRIAL: NCT03018392
Title: Fusion Rate and Clinical Outcomes Following 1 or 2 Level Open Transforaminal Lumbar Interbody Fusion for Degenerative Disc Disease With Novel 3-D Printed Titanium Cages With Pedicle Screw Fixation
Brief Title: Clinical and Radiological Evaluation of Patients With DDD Following TLIF With 3-D Printed Titanium Cage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bone and Joint Clinic of Baton Rouge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRITANIUM
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Intervertebral Disc Disease
MeSH Terms: conditions — Intervertebral disc disease

ARMS (1):
- Tritanium (Experimental): TLIF with Tritanium® PL cage and pedicle screw fixation
  Interventions: Device: Stryker Tritanium Spinal System

INTERVENTIONS:
Device: Stryker Tritanium Spinal System — open transforaminal lumbar interbody fusion (TLIF) utilizing the Stryker Tritanium cages with pedicle screw fixation according to instructions for use and package labeling for on-label indications

SUMMARY:
The purpose of this study is to evaluate the fusion rate and clinical outcomes at 1 year of 20 patients with degenerative disc disease who undergo a Transforaminal Lumbar Interbody Fusion (TLIF) with the Stryker Tritanium Spinal System. This is an on-label, post-market outcomes study to build on the body of long-term evidence for the device.

ELIGIBILITY:
Inclusion Criteria:

* Subject has one or more of the following diagnoses: degenerative disc disease (DDD) at one level or two contiguous levels from L2 to S1, and may also include up to Grade I spondylolisthesis at the involved level(s); degenerative scoliosis for which the Tritanium PL cage will be used as an adjunct to fusion
* Skeletally mature and ≥ 18 years old at time of enrollment
* Completed at least 6 months of non-operative therapy prior to surgery
* Willing and able to sign a study specific consent and comply with the requirements of the protocol including follow up visits and imaging.

Exclusion Criteria:

* 2 levels requiring surgical intervention
* Non-degenerative pathology including tumor, trauma, post-laminectomy kyphosis
* Psudeoarthrosis at the index level
* Previous fusion at the levels to be treated or at adjacent level
* Any abnormality present which affects the normal process of bone remodeling including, but not limited to, severe osteoporosis involving the spine, bone absorption, osteopenia, primary or metastatic tumors involving the spine, active infection at the site or certain metabolic disorders affecting osteogenesis.
* History of osteoporotic fracture
* History of an endocrine or metabolic disorder known to affect bone and mineral metabolism
* Inadequate tissue coverage over the operative site or taking medications that may interfere with bony/soft tissue healing including chronic steroid use
* Known allergy to titanium or cobalt chrome or may be sensitive to materials
* Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia
* Lumbar kyphosis- lumbar lordosis < 20°
* Degenerative scoliosis >20° OR any other pathology scoliosis (idiopathic, congenital, posttraumatic, iatrogenic)
* Active systemic infection or infection at the operative site
* Marked local inflammation
* Any open wounds
* Pregnant, or intends to become pregnant during the study
* Current smokers
* Subject is class 3 obese (BMI >40) or overweight and can produce loads on the spinal system which can lead to failure of the fixation of the device or to failure of the device itself
* Any mental or neuromuscular disorder which would create an unacceptable risk of fixation failure or complications in postoperative care
* Any neuromuscular deficit which places an unsafe load level on the device during the healing period
* Any other medical or surgical condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors, congenital abnormalities, elevation of sedimentation rate unexplained by other diseases, elevation of white blood cell count (WBC), or marked left shift in the WBC differential count.
* Any condition of senility, mental illness, or substance abuse.
* Involved in current spinal litigation that may interfere or influence patient self-assessment of function and pain
* Physical or mental condition that may interfere or influence patient self-assessment of function and pain.
* Incarcerated at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chambliss Harrod, MD, Principal Investigator — Bone and Joint Clinic of Baton Rouge

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tritanium
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tritanium
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (4)

OUTCOME MEASURES:

1. Primary Outcome: Fusion Rate
Description: Fusion status at 1 year post-operatively was graded as - fused (best outcome), progressing, or pseudoarthrosis (failed fusion)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanium
Number analyzed (Participants) | 20
Participants
  Fused | 19
  Pseudoarthrosis | 1
  Progressing | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tritanium
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tritanium (N=20)
Extension of fusion (Surgical and medical procedures) | 1 (1) — 1 subject had a locked pseudoarthrosis with progressive isthmic spondylolisthesis at an adjacent level. This necessitated an extension of fusion.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tritanium (N=20)
Cage Fracture (Product Issues) | 1 (1) — One incidental cage fracture in a setting of solid fusion was noted in the CT analysis. No intervention was necessary as the subject was doing well.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03018392/Prot_SAP_000.pdf